CLINICAL TRIAL: NCT03873389
Title: Evaluating the Effects of Ocrelizumab on the Circulating Metabolome in Multiple Sclerosis (MS)
Brief Title: Ocrelizumab Effects on the Metabolome in MS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00205181
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocrelizumab: All participants enrolled in the study. All participants will be receiving the treatment of interest (Ocrelizumab)
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Patients who are beginning this medication based on patient's treating physician's recommendation will be enrolled in the study.
  Other Names: Ocrevus

SUMMARY:
In this observational study, the investigators aim to recruit 50 patients over an 10-12 month period. The investigators will recruit patients with relapsing-remitting MS (based on 2017 McDonald Criteria) beginning treatment with ocrelizumab and fulfilling study inclusion and exclusion criteria. Participants recruited in this study will be participants in the Johns Hopkins MS Precision Medicine Center of Excellence bio-banking protocol which requires collection of serum and plasma at 6-monthly intervals and hence will have blood collection performed prior to Ocrevus start and then at 6, 12, 18 and 24 months following ocrelizumab initiation as part of the bio-banking protocol. All recruited participants will provide written informed consent.

The investigators will collect demographic and clinical characteristics at baseline and update these at follow-up visits. These will include disease duration, co-morbidities, relapses, treatment status and history. The investigators will also collect physiological variables - height and weight at each visit.

All recruited patients will return for follow up visits at 6,12, 18 and 24 months post-ocrelizumab initiation. At each visit patients will undergo the following evaluations - EDSS, MSFC, SDMT, fatigue scale (MFIS), quality of life measure (MS-QOL), depression scale (Beck depression inventory, 2nd version) and Block Food Frequency Questionnaire.

The investigators will then utilize plasma collected at the various time points to perform global metabolomics analysis. This will yield measures of various metabolites in the circulation, including amino acids and metabolites of the amino acids. The investigators will utilize this data to determine the change in the circulating metabolome produced by treatment with ocrelizumab.

Following this the investigators will assess changes in the various clinical measures collected - disability (EDSS, MSFC), cognition (SDMT), mood (BDI-II), fatigue (MFIS) and quality of life (MS-QOL) with Ocrelizumab treatment and correlate these with the changes noted in the metabolome. This approach will allow us to determine whether the metabolic changes are associated with/ could underlie the changes noted in clinical measures.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-75 years of age
* Diagnosis of relapsing remitting multiple sclerosis (RRMS) based on 2017 McDonald Criteria
* Initiating treatment with Ocrelizumab based on decision of the treating physician
* Able to return for visits every 6 months to Johns Hopkins MS Center

Exclusion Criteria:

* Presence of additional neuroinflammatory or neurodegenerative disorder
* Steroids within the past 30 days
* Other significant metabolic comorbidity - eg: uncontrolled hypothyroidism or diabetes
* Likely to switch therapy in the following year
* Previous treatment with rituximab or other chemotherapy agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients diagnosed with relapsing remitting multiple sclerosis between 18 and 75 years of age who are being started on ocrelizumab by the treating neurologist, are willing to return for visits every six months and do not have any other neurological disorder or significant metabolic comorbidity.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change in Global metabolomic profile | Baseline to 24 months
  Change in relative abundance of various metabolites, including amino acids and metabolites of the amino acids, in plasma measured using mass spectrometry

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale | Baseline to 24 months
  Change in level of disability as measured by a structured neurological examination resulting in the participants being rated on a scale from 1-10. Higher scores reflect greater physical disability.
Change in Multiple Sclerosis Functional Composite score | Baseline to 24 months
  Change in the multiple sclerosis functional composite which consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score (number of standard deviations away from mean of a normal population) with lower scores representing greater abnormality.
Change in Modified Fatigue Impact Scale score | Baseline to 24 months
  Change in scores on the modified fatigue impact scale which has 21 questions regarding the impact of fatigue on daily activities and scores range from 0-84. Higher scores reflect greater impact of fatigue on functioning.
Change in Multiple Sclerosis Quality of Life score | Baseline to 24 months.
  Change in physical and mental health scores as assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54) instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. Two summary scores - physical health and mental health - are derived from a weighted combination of scale scores. Higher scores suggest a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Bhargava, MBBS, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No